CLINICAL TRIAL: NCT01042600
Title: Rescue Surfactant for Respiratory Distress Syndrome (RDS) in Newborns: Comparing Efficacy of Delivery Via Laryngeal Mask Airway to Delivery by Endotracheal Intubation
Brief Title: Randomized Controlled Trial of Surfactant Delivery Via Laryngeal Mask Airway (LMA) Versus Endotracheal Intubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albany Medical College (Other)
Collaborators: ONY (Industry); LMA North America, Inc. (Industry)
Responsible Party: Principal Investigator, Joaquim M.B. Pinheiro, Professor of Pediatrics, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2599
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: Respiratory distress syndrome; Surfactant; Tracheal intubation; Laryngeal mask airway; Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Respiratory Distress Syndrome | interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endotracheal intubation (Active Comparator): Endotracheal tube insertion for surfactant administration, following morphine and atropine pre-medication
  Interventions: Device: Endotracheal tube insertion
- Laryngeal mask airway (Experimental): Laryngeal mask airway insertion for surfactant administration, following atropine pre-medication
  Interventions: Device: Laryngeal mask airway insertion

INTERVENTIONS:
Device: Endotracheal tube insertion — Endotracheal tube insertion after premedication with atropine (0.02 mg/kg) and morphine (0.1 mg/kg)
  Arms: Endotracheal intubation
Device: Laryngeal mask airway insertion — Laryngeal mask airway insertion after premedication with atropine (0.02 mg/kg)
  Other Names: LMA North America
  Arms: Laryngeal mask airway

SUMMARY:
In this study, newborn babies with respiratory distress syndrome (RDS), receiving oxygen via nasal CPAP, and needing surfactant treatment will be randomized to standard delivery of surfactant via and endotracheal tube airway(inserted after pre-medication for pain), or to surfactant delivery via laryngeal mask airway (LMA). The intent is to remove the airways and return babies to nasal CPAP, after surfactant is given. The primary outcome measure is the rate of failure of initial surfactant therapy. Standardized failure criteria are reached: a) early, if the baby is unable to be placed back on CPAP (needs mechanical ventilation) or, b) late, if the baby requires retreatment with surfactant within 8 hours or more than 2 doses of surfactant.

The objective of this protocol is to reduce the need for endotracheal intubation and mechanical ventilation in preterm neonates with RDS needing rescue surfactant therapy by instilling surfactant though an LMA, while achieving comparable efficacy of surfactant treatment.

The hypothesis is that surfactant treatment through an LMA will decrease the proportion of babies with RDS who require mechanical ventilation or subsequent intubation, when compared with standard surfactant treatment following sedation and endotracheal intubation.

DETAILED DESCRIPTION:
Respiratory Distress Syndrome (RDS) due to deficiency of lung surfactant is common in preterm newborns. Early treatment with surfactant improves oxygenation, reduces the need for subsequent mechanical ventilation, decreases the incidence of pulmonary air leaks and chronic lung disease and it also reduces mortality in extremely premature newborns. Optimal treatment of RDS includes surfactant therapy and avoidance of invasive mechanical ventilation by using nasal continuous positive airway pressure (NCPAP). The current standard method of surfactant delivery requires tracheal intubation and at least brief positive-pressure ventilation. Tracheal intubation causes pain and leads to vagal-mediated physiologic instability in neonates; therefore, premedication with morphine and atropine is routinely practiced in our setting. However, premedication with morphine often increases respiratory depression, requiring sustained mechanical ventilation. The Laryngeal Mask Airway (LMA) is a commercially available, less invasive artificial airway that does not need to be inserted into the trachea; it is FDA-approved for use in neonates, and preliminary data suggest that it can be used for surfactant administration.

The main objective of this study protocol is reduce the need for endotracheal intubation and mechanical ventilation in preterm neonates with mild to moderate RDS needing rescue surfactant therapy by instilling surfactant though an LMA. A second objective is to compare the efficacy of surfactant administered via LMA versus endotracheal tube (ETT) in decreasing the severity of RDS. Additionally, we will evaluate the safety of surfactant administration via LMA.

The primary hypothesis is that surfactant treatment via the LMA approach will decrease the proportion of babies with RDS who require mechanical ventilation or subsequent intubation, when compared with standard surfactant as administered to the ETT group.

This randomized controlled trial will include babies with mild-to-moderate RDS, between 4 to 48 hours of age, with gestational age 29 0/7 to 36 6/7 weeks, treated with NCPAP ≥ 5 cm H2O and FiO2 between 0.30 and 0.60 for at least 2 hours to maintain SpO2 88-95%, and informed consent. Exclusion criteria are weight < 1000 g, airway anomalies, pulmonary air leaks, and craniofacial and cardiothoracic malformations.

After informed consent is obtained, babies are randomly assigned (from sealed, opaque, consecutively numbered envelopes), to the "ETT" or "LMA". The "ETT" group is managed according to our current practice of surfactant therapy (endotracheal intubation following premedication with atropine + morphine), whereas the "LMA" group will be pre-medicated with atropine before LMA insertion for surfactant administration.

Both groups will receive Infasurf (3mL/kg) instilled in 2 aliquots via their respective airway, followed by PPV for at least 5 minutes. The artificial airway will be removed and the patient returned to NCPAP by 15 minutes, if spontaneous respirations are adequate. Indications for surfactant re-dosing and mechanical ventilation will be equivalent for both groups.

Babies will continue or initiate assisted ventilation via ETT if any of the following occurs:

* Persistent apnea;
* Severe retractions;
* Inability to wean FiO2 < 60%

Criteria for re-dosing with surfactant:

1. Within 8 hours after first dose of surfactant (early re-dosing):

   * FiO2 20% higher than the baseline FiO2, after excluding other obvious causes of respiratory insufficiency such as pneumothorax.

   If early re-dosing of surfactant is needed in patients of either group, the dose will be administered via ETT (i.e., LMA patients will be intubated, and will receive the dose of surfactant via ETT)
2. Beyond 8 hours of the first dose of surfactant (late re-dosing):

   * FiO2 is ≥ 60%, or;
   * FiO2is ≥ 30% associated with worsening clinical signs of RDS.

If late re-dosing is needed in patients of the LMA group, use of the LMA is permitted for the second dose. In the ETT group, all doses are given via the ETT.

Primary Outcome Measures:

Rate of failure of early surfactant rescue therapy in the 2 groups, using the following criteria to differentiate early from late failure:

* Criteria for early failure (within 1 hour):

  1. The need of mechanical ventilation within 1 hour of surfactant therapy.
  2. Use of Narcan to avoid mechanical ventilation after surfactant therapy.
* Criteria for late failure (beyond 1 hour):

  1. Sustained FiO2 > 0.60 to maintain target SpO2
  2. Second dose of surfactant within 8 hours after the first dose.
  3. More than 2 doses of surfactant.

Babies will have FiO2 adjusted to maintain SpO2 88-95%, per current practice. Other aspects of weaning ventilatory support will be managed by clinicians' preference.

ELIGIBILITY:
Inclusion Criteria:

* Mild-to-moderate RDS
* Postnatal age 4 to 48 hours
* Gestational age 29 0/7 to 36 6/7 weeks
* Treated with nasal CPAP ≥ 5 cm H2O and FiO2 between 0.30 and 0.60 for at least 2 hours to maintain SpO2 88-95%
* Informed consent

Exclusion Criteria:

* Weight < 1000 g
* Airway anomalies
* Pulmonary air leaks
* Craniofacial or cardiothoracic malformations

Ages: 4 Hours to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2009-12; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim M Pinheiro, MD, MPH, Principal Investigator — Albany Medical College; Querube Santana, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant excluded and removed from study after randomization due to ineligibility (pre-existing pneumothorax)
Groups:
- Endotracheal Intubation: Endotracheal intubation for surfactant administration, following morphine and atropine pre-medication
  Endotracheal tube insertion: Endotracheal tube insertion after premedication with atropine (0.02 mg/kg) and morphine (0.1 mg/kg)
Period: Overall Study
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Started | 31 | 30
Completed | 30 | 30
Not Completed | 1 | 0
Not completed — Ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Population: Single ineligible patient excluded in the endotracheal intubation group
Groups:
- Total: Total of all reporting groups
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Customized [Number; unit: participants]
  Gestational age <33 weeks | 18 | 11 | 29
  Gestational age >=33 weeks | 13 | 19 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 18 | 21 | 39

OUTCOME MEASURES:

1. Primary Outcome: Rate of Failure of Surfactant Therapy, Either Early (Need for Mechanical Ventilation Within 1 Hour), or Late (FiO2 > 0.60 to Maintain Target SpO2, or Second Dose of Surfactant Within 8 Hours, or Needing More Than 2 Doses of Surfactant).
Time Frame: 96 hours
Measure: Number; unit: participants
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 30 | 30
participants | 23 | 9

2. Secondary Outcome: Number of Surfactant Doses
Description: Mean number of surfactant doses
Time Frame: 96 hr
Measure: Mean (Standard Deviation); unit: mean doses
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 30 | 30
mean doses | 1.3 (.6) | 1.8 (1.0)

3. Secondary Outcome: Days on Assisted Ventilation
Description: Days on any respiratory support
Time Frame: 2 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 30 | 30
days | 11 [7 to 21] | 8.5 [6 to 22]

4. Secondary Outcome: Days on Supplemental Oxygen
Time Frame: 2 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 30 | 30
days | 10 [6 to 20] | 7.5 [4 to 19]

5. Secondary Outcome: Rate of Pneumothorax
Time Frame: 96 hrs
Measure: Number; unit: percentage of participants
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 30 | 30
percentage of participants | 13 | 20

6. Secondary Outcome: Rate of BPD (O2 Dependence at the Later of 28 Days of Age or 36 Weeks Postmenstrual Age)
Time Frame: 2 months
Measure: Number; unit: percentage of participants
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 30 | 30
percentage of participants | 7 | 10

7. Secondary Outcome: Complications During Insertion of LMA
Description: LMA insertion complications (e.g. trauma, failure of insertion)
Time Frame: 96 hrs
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

8. Secondary Outcome: Mortality Rate
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 30 | 30
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 10/30 | 7/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endotracheal Intubation (N=30) | Laryngeal Mask Airway (N=30)
Bradycardia (Cardiac disorders) | 6 (6) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) — Pneumothorax after randomization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No